CLINICAL TRIAL: NCT00424489
Title: Hematopoietic Stem Cell Therapy for Patients With Refractory Myasthenia Gravis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled for more than two years. No plan to continue study.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myasthenia Gravis Auto 2002
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Myasthenia Gravis
Keywords: Refractory Myasthenia Gravis; Autologous Stem Cell Transplantation; Cyclophosphamide and ATG
MeSH Terms: conditions — Myasthenia Gravis | interventions — Hematopoietic Stem Cell Transplantation; Cyclophosphamide; thymoglobulin; Mesna; Methylprednisolone; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Autologous Hematopoietic Stem Cell Transplantation will be performed after conditioning
  Interventions: Biological: Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: ATG (rabbit); Drug: Mesna; Drug: Methylprednisolone; Drug: G-CSF

INTERVENTIONS:
Biological: Hematopoietic Stem Cell Transplantation — Autologous Hematopoietic Stem Cell Transplantation
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: ATG (rabbit)
Drug: Mesna
Drug: Methylprednisolone
Drug: G-CSF

SUMMARY:
MG may be neonatal, congenital, or autoimmune. Neonatal MG arises from transplacental transfer of ACh receptor antibodies from a mother with autoimmune MG to the fetus. Neonatal MG resolves with post delivery clearance of maternal antibodies. Congenital MG results from a genetic defect in the ACh receptor. Patients with congenital MG do not have ACh receptor antibodies. Both neonatal and congenital MG are excluded from this study. Autoimmune MG, which is the most common form of MG, affects approximately 25,000 Americans. Like most autoimmune diseases, it is associated with particular HLA genotypes, has a female predominance, and environmental factors involved in breaking tolerance to the ACh receptor are unknown. Patients with refractory and severe autoimmune MG will be considered candidates for this study.

The purpose of this study is to assess the toxicity/feasibility (phase I) of autologous hematopoietic stem cell transplantation for refractory myasthenia gravis.

DETAILED DESCRIPTION:
There will be no randomization in this study. All subjects who are determined to be eligible for the study treatment will receive high dose cyclophosphamide and ATG followed by infusion of autologous peripheral blood stem cells. The procedures the subject will undergo are as follows:

1. Physician visit to determine potential eligibility for the study. Subjects will be evaluated by a transplant physician and a neurologist. They will have a complete physical examination and will provide a full medical history at these visits. The study will be described in detail by the transplant physician and nurse and the consent form will be provided to be taken home to read.
2. Insurance verification. Subjects who remain interested in pursuing the study treatment and who have refractory myasthenia gravis will proceed to the insurance verification phase. Third party payment or self-pay must be verified before subjects can proceed.
3. Consent form. Prior to proceeding, the appropriate signatures will be obtained on the consent form. Subjects will be given an opportunity to ask further questions of the attending physician and transplant nurse prior to signing the consent form.
4. Pre-transplant testing. To determine final eligibility for the study, subjects will undergo a series of tests/procedures. These include: CXR; electrocardiogram; MUGA or echocardiogram; pulmonary function test; CT scan of the sinuses; CT scan of the chest to r/o thymoma; dental examination; urinalysis; and blood testing to include CBC, chemistries, liver and kidney function tests, coagulation studies, viral studies and, for females, a pregnancy test. All pre-transplant testing is routine medical testing done to verify diagnosis and to insure adequate organ function and absence of viral illnesses which would preclude a safe transplant course.
5. Autologous peripheral blood stem cell collection. Subjects who are proceeding to transplant will undergo a routine procedure for the mobilization and collection of peripheral blood stem cells. This includes the administration of IV cyclophosphamide, given as an inpatient requiring an overnight stay, followed by the subcutaneous administration of G-CSF, to be self-administered as an outpatient. Approximately ten days after the administration of IV cyclophosphamide, the peripheral blood stem cells will be collected as an outpatient in the Blood Center. A pheresis catheter will be placed for this purpose on the first day of leukopheresis. Leukopheresis will be continued on a daily basis until an adequate number of peripheral blood stem cells have been collected (a maximum of four leukophereses may be performed). G-CSF will continue to be administered until leukopheresis is completed. The pheresis catheter will be discontinued when stem cell harvesting is completed. Processed cells will be frozen and stored until they are reinfused after the conditioning regimen.
6. PICC line placement. Subjects will have a double lumen PICC line placed prior to the administration of study treatment for the administration of chemotherapy, IV fluids, blood products and the withdrawal of blood samples. The placement of a PICC line is a routine medical procedure.
7. Study treatment. Subjects will undergo conditioning which will include four days of intravenous high dose cyclophosphamide and three days of intravenous anti-thymocyte globulin (ATG). Both cyclophosphamide and ATG are common immune suppressive agents. The previously collected peripheral blood stem cells will be reinfused following the completion of the conditioning regimen.
8. Post-treatment follow-up. Subjects will have a history and physical by the transplant physician and neurologist at 3 months, 6 months, 12 months, and yearly for 5 years. In addition, routine urinalysis and blood testing will be performed at these same intervals to include CBC, chemistries, kidney and liver function tests.

ELIGIBILITY:
Inclusion Criteria (Patients must fulfill all of the following)

1. Established diagnosis of myasthenia gravis defined as clinical evidence of muscle weakness and fatigue ability and supported, an abnormal EMG-NCV repetitive nerve stimulation (or single-fiber EMG) or Lambert-Eaton Myasthenic Syndrome without evidence of malignancy.
2. Ages 15-65 years.
3. Positive antibody preferred (anti-AchR, MuSK, voltage gated calcium channel, anti-striational).
4. Failure of thymectomy (except for Lambert-Eaton Myasthenic Syndrome).
5. Failure anticholinesterase therapy, corticosteroids, and at least two of the following: azathioprine, cyclosporin, CellCept, cyclophosphamide, plasma exchange, or IVIG. Failure is defined as at least 6 months of the above drug therapy and an Osserman score of IIB, III, or IV and not clinically improving.

And at least one of the following:

1. History of myasthenia crises (requiring mechanical ventilation) despite thymectomy and immunosuppressive therapy.
2. Hospitalized or on ventilator support for myasthenia gravis within the last 18 months despite thymectomy and immunosuppressive therapy.
3. Inability to maintain nutrition due to muscle weakness.
4. A Karnofsky performance status of 70% or less (may or may not be able to care for self, but unable to carry on normal activity or unable to do active work).

Exclusion Criteria

1. Significant end organ damage such as:

   1. LVEF <40% or deterioration of LVEF during exercise test on MUGA or echocardiogram.
   2. Untreated life-threatening arrhythmia, active ischemic heart disease or heart failure.
   3. DLCO < 40% of predicted value.
   4. Serum creatinine > 2.5 mg/dl.
   5. Liver cirrhosis, transaminases >3x of normal limits, or bilirubin >2.0 unless due to Gilberts disease.
2. HIV positive.
3. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
4. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer, will be considered on an individual basis.
5. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
7. Inability to give informed consent
8. Congenital myasthenia gravis
9. Neonatal myasthenia gravis
10. Osserman grade 1 or 2
11. Pure red cell aplasia
12. Any patient on insulin

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University and Northwestern Memorial Hospital
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 9
Completed | 6
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.22 (16.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival
Time Frame: Up to 5 years
Population: Survival both treatment related and non-treatment related
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 9
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=9)
Methicillin-Resistant Staphylococcus Aureus (MRSA) (Infections and infestations) | 1 (1) — One patient with prior splenectomy and thymectomy died of sepsis bacteremia.
Insulin induced hypoglycemia (Endocrine disorders) | 1 (9) — One known diabetic on tight insulin control died of insulin overdose.
High Grade Lymphoma (Blood and lymphatic system disorders) | 1 (1) — One participant died of late lymphoma.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=9)
GR+ bacteriemia (Infections and infestations) | 1 (1) — One patient developed pneumonia, resolved with antibiotics.
pneumonia (Infections and infestations) | 1 (1) — One patient with post transplant pneumonia resolved with antibiotics.
Seizure (Nervous system disorders) | 1 (1) — One participant was hospitalized after having seizure. The cause was idiopathic and workup was negative except for pituitary cyst, treated with Keppra with no further seizures.
bowl obstruction (Gastrointestinal disorders) | 1 (1) — One patient hospitalized for bowl obstruction that resolved without surgical intervention.

LIMITATIONS AND CAVEATS:
Small numbers of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes